CLINICAL TRIAL: NCT07305766
Title: Construction and Preliminary Application of Evidence-Based Nursing Protocol for Oral Mucositis Related to Tumor Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Yutong XU, Master, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: No. PUMCSON-2023-26
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Oral Mucositis (Ulcerative) Due to Antineoplastic Therapy
Keywords: Evidence-Based Nursing Protocol; Oral Mucositis
MeSH Terms: conditions — Stomatitis; Ulcer | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): In addition to providing patients with oral hygiene education (brushing teeth twice daily and rinsing with water after meals) and administering symptomatic treatment as prescribed, during their outpatient infusion visits, nurses will deliver evidence-based nursing interventions for cancer therapy-related oral mucositis through face-to-face education and guidance. Following discharge, patients will receive weekly online follow-up visits to enhance adherence to the protocol. Additionally, patients will be monitored for any adverse reactions or intolerance symptoms-such as nausea and vomiting-during the implementation of the evidence-based oral mucositis care regimen.
  Interventions: Behavioral: Conventional nursing measures
- Intervention group (Experimental): In addition to providing patients with oral hygiene education (brushing teeth twice daily and rinsing with water after meals) and administering symptomatic treatment as prescribed, during their outpatient infusion visits, nurses will deliver evidence-based nursing interventions for cancer therapy-related oral mucositis through face-to-face education and guidance. Following discharge, patients will receive weekly online follow-up visits to enhance adherence to the protocol. Additionally, patients will be monitored for any adverse reactions or intolerance symptoms-such as nausea and vomiting-during the implementation of the evidence-based oral mucositis care regimen.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — In addition to providing patients with oral hygiene education (brushing teeth twice daily and rinsing with water after meals) and administering symptomatic treatment as prescribed, during their outpatient infusion visits, nurses will deliver evidence-based nursing interventions for cancer therapy-related oral mucositis through face-to-face education and guidance. Following discharge, patients will receive weekly online follow-up visits to enhance adherence to the protocol. Additionally, patients will be monitored for any adverse reactions or intolerance symptoms-such as nausea and vomiting-during the implementation of the evidence-based oral mucositis care regimen.
  Arms: Intervention group
Behavioral: Conventional nursing measures — Conventional nursing measures were provided, entailing patient education on oral care (brushing twice daily and rinsing with plain water postprandially), as well as symptom management according to established protocols.
  Other Names: Control group
  Arms: Control group

SUMMARY:
Describe the incidence and influencing factors of cancer therapy-related oral mucositis. Based on evidence-based practice, develop a standardized nursing protocol for cancer therapy-related oral mucositis that aligns with China's national context and demonstrates strong clinical feasibility, and establish a clinical management pathway for cancer therapy-related oral mucositis. Validate the implementability of the standardized nursing protocol, and evaluate its clinical effectiveness and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed cancer diagnosis who are aware of their condition.
* Patients currently undergoing non-surgical treatments such as chemotherapy, radiotherapy, immunotherapy, or targeted therapy.
* Patients who voluntarily agree to participate in this study and provide informed consent.

Exclusion Criteria:

* Patients with autoimmune diseases;
* Patients with primary or metastatic oral or lip cancer.;
* Patients who are participating in other intervention studies.;
* Swallowing problems existed in patients with Kubota drinking test > level 3;
* Coma or inability to open mouth, difficulty cooperating with the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of oral mucositis | One treatment cycle (21days)
  WHO Oral Mucositis Assessment Scale

SECONDARY OUTCOMES:
Oral Condition Assessment | One treatment cycle (21days)
  Oral Assessment Guide
Salivary pH | One treatment cycle (21days)
  Salivary pH was measured using pH test paper. Prior to testing, participants were required to fast (including no food or water) for one hour and to avoid activities that might alter salivary composition, such as using mouthwash, brushing teeth, smoking, or chewing gum. After one hour, a saliva sample was collected. Using a dropper, a sample was placed onto the pH test paper until it was fully saturated. After waiting for 10 seconds, the color change was compared against a standard color chart. Normal salivary pH typically falls within the range of 6.6 to 7.1, with a lower pH value indicating higher salivary acidity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Published on ResMan (http://www.medresman.org.cn/)
Supporting Information: Study Protocol
Time Frame: Publication date: January 30, 2028

REFERENCES:
- [Result] Xu Y, Wang J, Zhang Y, Guo Z, Zhang W, Zhang S, Shi W, Ma W. Occurrence and Influencing Factors of Oral Mucositis in Patients With Cancer: A Cross-Sectional Study in China. Oncol Nurs Forum. 2025 Oct 20;52(6):460-472. doi: 10.1188/25.ONF.460-472. PMID 41123400